CLINICAL TRIAL: NCT03767413
Title: The Effects of Mental Practice Combined With Proprioceptive Neuromuscular Facilitation on Muscle Strength of Upper Limb and Hand Grip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Wafaa Mahmoud Amin, Principal investigator, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 8810025277
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Motor Activity; Physical Activity; Neuromuscu
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: There are two group of subjects: PNF group will receive only PNF training PNFMP group: will receive PNF training and mental pracice technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF group (Active Comparator): It will be consisted of 15 -25 healthy subjects receiving only proprioceptive nueromuscular facilitation training for 5 weeks with 17 days follow up after completion of program.
  Interventions: Procedure: PNF
- PNFMP (Experimental): It will be consisted of 15 -25 healthy subjects receiving proprioceptive nueromuscular facilitation training and mental practice technique for 5 weeks with 17 days follow up after completion of program.
  Interventions: Procedure: PNFMP

INTERVENTIONS:
Procedure: PNF — proprioceptive neuromuscular facilitation training
  Arms: PNF group
Procedure: PNFMP — proprioceptive neuromuscular facilitation training and mental practice technique
  Arms: PNFMP

SUMMARY:
Influence of mental practice and proprioceptive neuromuscular facilitation on muscle strength of upper limb and hand grip will be measured in 30 to 50 healthy students with right dominant hand, Their age will be ranged from 18 to 26 years old. Subjects will randomly assigned to either proprioceptive neuromuscular facilitation (PNF) group or proprioceptive neuromuscular facilitation with mental practice (PNFMP) group.

DETAILED DESCRIPTION:
PNF group: 15 - 25 individuals, these subjects will receive only PNF training. PNFMP: 15 individuals, these subjects will receive PNF training with MP. Training program will be conducted for every group for 5 weeks with 3 sessions x 30 min per week. Electromyography (EMG) device will be used to measure the electrical activity of muscles using surface electrodes. Hydraulic hand dynamometer will be used to measure hand grip strength.

ELIGIBILITY:
Inclusion Criteria:

1. The participant will be right-handed.
2. Previously untrained subjects.
3. Absence of a prior injury of the hand or arm

Exclusion Criteria:

1. History of a neurological disease.
2. History of musculoskeletal injury of upper limb.
3. Unstable medical condition

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Shoulder joint strength | 6 minutes
  electromyography device will be used to measure the electrical activity of the muscle
Elbow joint strength | 6 minutes
  electromyography device will be used to measure the electrical activity of the muscle
Strength of hand grip | 15 minutes
  Hand held dynamometer will be used to measure the strength of the hand grip

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
there is no plan